CLINICAL TRIAL: NCT04786444
Title: A Randomized, Double-Blinded Phase 3 Study to Demonstrate Lot-to-Lot Consistency of Three Lots of a Live-Attenuated Chikungunya Virus Vaccine Candidate (VLA1553) in Healthy Adults Aged 18 to 45 Years
Brief Title: Study to Demonstrate Consistency of Three Lots of a Live-attenuated Chikungunya Virus Vaccine Candidate in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA1553-302
Record Dates: First submitted 2021-02-22; First posted 2021-03-08 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chikungunya Virus Infection
Keywords: VLA1553; Chikungunya Virus Infection; CHIKV; Live-attenuated Chikungunya virus vaccine
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VLA1553 Lot 1 (Active Comparator)
  Interventions: Biological: Biological Vaccine VLA1553
- VLA1553 Lot 2 (Active Comparator)
  Interventions: Biological: Biological Vaccine VLA1553
- VLA1553 Lot 3 (Active Comparator)
  Interventions: Biological: Biological Vaccine VLA1553

INTERVENTIONS:
Biological: Biological Vaccine VLA1553 — Single intramuscular vaccination on Day 1 with one of three Lots of VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate

SUMMARY:
This was a prospective, randomized, double-blinded, multicenter Phase 3 clinical study investigating three Lots of VLA1553 at the final dose. Overall 409 healthy subjects aged 18 to 45 years were randomized into the study.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blinded, multicenter Phase 3 clinical study investigating three Lots of VLA1553. Overall 409 healthy subjects aged 18 to 45 years were randomized into the study, approximately136 subjects per VLA1553 Lot. Subjects were block-randomized in a 1:1:1 ratio into the three study arms to receive one of three Lots of VLA1553 as a single i.m. vaccination. The primary objective was to demonstrate Lot-to-Lot manufacturing consistency of VLA1553 28 days following the single vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years of age on the Day of screening
2. Able to provide informed consent
3. Generally healthy as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests
4. For women of childbearing potential:

   1. practiced an adequate method of contraception during 30 days before screening
   2. negative serum or urine pregnancy test at screening or vaccination, respectively
   3. agreed to employ adequate birth control measures for the first three months post-vaccination.

Exclusion Criteria:

1. CHIKV infection in the past (self-reported), including suspected CHIKV infection; was taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or had participated in a clinical study involving an investigational CHIKV vaccine
2. Acute or recent infection (and not symptom-free in the week prior to screening)
3. Tested positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
4. Received another live virus vaccine within 28 days or inactivated vaccine within 14 days prior to vaccination in this study or plans to receive a vaccine within 28 days or 14 days after vaccination, respectively
5. Abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the study
6. Medical history of or currently had acute or progressive, unstable or uncontrolled clinical conditions that posed a risk for participation in the study
7. History of immune-mediated or clinically relevant arthritis / arthralgia
8. History of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there had been surgical excision or treatment more than 5 years ago that was considered to have achieved a cure, the subject could be enrolled.
9. Known or suspected defect of the immune system, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to vaccination.
10. History of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications)
11. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws
12. Pregnant, had plans to become pregnant during the first three months post-vaccination or lactating at the time of enrollment
13. Donation of blood, blood fractions or plasma within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or planned to donate blood or use blood products until Day 180 of the study
14. Rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating
15. Known or suspected problem with alcohol or drug abuse as determined by the Investigator
16. Any condition that, in the opinion of the Investigator, could compromise the subjects well-being, could interfere with evaluation of study endpoints, or could limit the subject's ability to complete the study;
17. Committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities)
18. Participation in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study
19. Member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 409 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (12):
- United States (12):
  - AMR Miami, Coral Gables, Florida
  - AMR Fort Myers, Fort Myers, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - AMR Wichita West, Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Walter Reed Amy Institute of Research, Silver Spring, Maryland
  - Alliance for Multispecialty Research (AMR), Kansas City, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - AMR Knoxville, Knoxville, Tennessee
  - Dynamed Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Started | 136 | 137 | 135
Completed | 121 | 120 | 123
Not Completed | 15 | 17 | 12
Not completed — Withdrawal by Subject | 4 | 7 | 2
Not completed — Lost to Follow-up | 11 | 9 | 10
Not completed — Subject would like to become pregnant | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3 | Total
Number analyzed (Participants) | 136 | 137 | 135 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (7.03) | 33.2 (7.78) | 33.2 (7.43) | 33.2 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 72 | 223
  Male | 61 | 61 | 63 | 185
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American, Indian or Alaska Native | 4 | 1 | 0 | 5
  Asian | 6 | 5 | 7 | 18
  Black or African American | 21 | 22 | 19 | 62
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  White | 103 | 106 | 106 | 315
  Other | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of CHIKV-specific Neutralizing Antibodies as Determined by Microneutralization (μPRNT) Assay in Subjects Who Tested Negative for CHIKV Antibodies at Baseline
Time Frame: On Day 29 after single vaccination
Population: The Per-Protocol population used for immunogenicity analyses, is based on participants without major protocol deviations that could impact the immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 122 | 118 | 122
Geometric Mean Titer | 2556.7 [2055.63 to 3179.80] | 2767.7 [2310.25 to 3315.65] | 2613.7 [2128.06 to 3210.17]

2. Secondary Outcome: Immune Response as Measured by CHIKV-specific Neutralizing Antibody Titers
Time Frame: on Day 8, 85 and Month 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 121 | 118 | 122
Geometric Mean Titer
  Visit 2 - Day 8: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8 | 13.0 [11.72 to 14.38] | 12.0 [11.04 to 13.03] | 11.4 [10.52 to 12.40]
  Visit 4 - Day 85: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85 | 832.3 [696.51 to 994.59] | 829.0 [688.88 to 997.51] | 875.8 [730.45 to 1050.12]
  Visit 5 - Day 180: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180 | 666.4 [546.33 to 812.97] | 777.6 [663.40 to 911.43] | 688.3 [573.46 to 826.25]

3. Secondary Outcome: Proportion of Subjects With Seroprotective Levels for Baseline Negative Subjects
Time Frame: on Day 8, 29, 85 and Month 6
Population: The Per-Protocol population used for immunogenicity analyses, is based on participants who have available Day 1 and Day 29 samples and without major protocol deviations that could impact the immune response
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 122 | 118 | 122
Participants
  Visit 2 - Day 8: number analyzed (Participants) | 110 | 110 | 111
  Visit 2 - Day 8 | 0 | 0 | 0
  Visit 3 - Day 29: number analyzed (Participants) | 120 | 116 | 120
  Visit 3 - Day 29 | 117 | 114 | 117
  Visit 4 - Day 85: number analyzed (Participants) | 108 | 107 | 115
  Visit 4 - Day 85 | 106 | 104 | 111
  Visit 5 - Day 180: number analyzed (Participants) | 109 | 108 | 112
  Visit 5 - Day 180 | 103 | 106 | 107

4. Secondary Outcome: Proportion of Subjects With Seroconversion
Time Frame: on Day 29, Day 85 and Month 6
Population: At the specified time point the number of subjects with non-missing titers is stated.
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 122 | 118 | 122
Participants
  Visit 3 - Day 29 | 118 | 116 | 119
  Visit 4 - Day 85: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85 | 107 | 106 | 115
  Visit 5 - Day 180: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180 | 107 | 108 | 112

5. Secondary Outcome: Fold Increase of CHIKV-specific Neutralizing Antibody Titers Compared to Baseline
Time Frame: on Day 8, 29, 85 and Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Fold increase
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 122 | 118 | 122
Fold increase
  Visit 2 - Day 8: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8 | 1.58 (1.570) | 1.37 (1.048) | 1.32 (1.460)
  Visit 3 - Day 29 | 379.56 (319.179) | 371.37 (294.164) | 399.91 (523.539)
  Visit 4 - Day 85: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85 | 110.92 (79.788) | 109.81 (76.375) | 123.20 (100.725)
  Visit 5 - Day 180: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180 | 96.20 (79.639) | 98.57 (71.635) | 97.24 (83.274)

6. Secondary Outcome: Proportion of Subjects Reaching an at Least 4-fold, 8-fold, 16-fold or 64-fold Increase in CHIKV-specific Neutralizing Antibody Titer Compared to Baseline
Time Frame: up to Month 6
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 122 | 118 | 122
Participants
  Visit 2 - Day 8: subjects reaching 4-fold increase: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8: subjects reaching 4-fold increase | 8 | 6 | 3
  Visit 2 - Day 8: subjects reaching 8-fold increase: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8: subjects reaching 8-fold increase | 1 | 0 | 1
  Visit 2 - Day 8: subjects reaching 16-fold increase: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8: subjects reaching 16-fold increase | 0 | 0 | 0
  Visit 2 - Day 8: subjects reaching 64-fold increase: number analyzed (Participants) | 112 | 112 | 113
  Visit 2 - Day 8: subjects reaching 64-fold increase | 0 | 0 | 0
  Visit 3 - Day 29: subjects reaching 4-fold increase | 118 | 116 | 119
  Visit 3 - Day 29: subjects reaching 8-fold increase | 118 | 116 | 119
  Visit 3 - Day 29: subjects reaching 16-fold increase | 117 | 116 | 119
  Visit 3 - Day 29: subjects reaching 64-fold increase | 116 | 116 | 116
  Visit 4 - Day 85: subjects reaching 4-fold increase: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85: subjects reaching 4-fold increase | 107 | 106 | 115
  Visit 4 - Day 85: subjects reaching 8-fold increase: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85: subjects reaching 8-fold increase | 107 | 106 | 114
  Visit 4 - Day 85: subjects reaching 16-fold increase: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85: subjects reaching 16-fold increase | 107 | 106 | 113
  Visit 4 - Day 85: subjects reaching 64-fold increase: number analyzed (Participants) | 110 | 109 | 117
  Visit 4 - Day 85: subjects reaching 64-fold increase | 75 | 71 | 77
  Visit 5 - Day 180: subjects reaching 4-fold increase: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180: subjects reaching 4-fold increase | 107 | 108 | 112
  Visit 5 - Day 180: subjects reaching 8-fold increase: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180: subjects reaching 8-fold increase | 107 | 108 | 110
  Visit 5 - Day 180: subjects reaching 16-fold increase: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180: subjects reaching 16-fold increase | 103 | 108 | 109
  Visit 5 - Day 180: subjects reaching 64-fold increase: number analyzed (Participants) | 111 | 110 | 114
  Visit 5 - Day 180: subjects reaching 64-fold increase | 69 | 69 | 64

7. Secondary Outcome: Frequency of Solicited Injection Site
Time Frame: 10 days post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  number of subjects experiencing any solicited injection site adverse events | 23 | 30 | 26
  Tenderness | 19 | 22 | 17
  Pain | 7 | 10 | 9
  Erythema/Redness | 4 | 2 | 5
  Induration | 3 | 1 | 3
  Swelling | 2 | 0 | 2

8. Secondary Outcome: Frequency of Solicited Systemic Reactions
Time Frame: 10 days post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  number of subjects experiencing any solicited systemic adverse events | 73 | 78 | 82
  Fatigue | 53 | 49 | 53
  Headache | 49 | 42 | 55
  Myalgia | 31 | 35 | 30
  Arthralgia | 19 | 21 | 23
  Nausea | 16 | 20 | 17
  Fever | 16 | 18 | 18
  Rash | 1 | 6 | 6
  Vomiting | 2 | 6 | 2

9. Secondary Outcome: Severity of Solicited Injection Site
Time Frame: 10 days post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  Mild | 21 | 29 | 26
  Moderate | 2 | 1 | 0
  Severe | 0 | 0 | 0

10. Secondary Outcome: Severity of Solicited Systemic Reactions
Time Frame: 10 days post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  Mild | 56 | 60 | 61
  Moderate | 12 | 15 | 18
  Severe | 5 | 3 | 3

11. Secondary Outcome: Severity of Unsolicited Adverse Events (AEs) Within 28 Days Post-vaccination
Time Frame: up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  Mild | 25 | 17 | 32
  Moderate | 10 | 5 | 10
  Severe | 3 | 0 | 0

12. Secondary Outcome: Frequency of Unsolicited Adverse Events (AEs) Within 28 Days Post-vaccination
Time Frame: up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants | 38 | 22 | 42

13. Secondary Outcome: Severity of Any Adverse Event During the Entire Study Period
Time Frame: up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  Mild | 64 | 66 | 61
  Moderate | 26 | 27 | 36
  Severe | 8 | 4 | 4

14. Secondary Outcome: Frequency of Any Adverse Event During the Entire Study Period
Time Frame: up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants | 98 | 97 | 101

15. Secondary Outcome: Frequency of Any Serious Adverse Event (SAE) During the Entire Study Period
Time Frame: up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants | 3 | 2 | 0

16. Secondary Outcome: Severity of Any Adverse Event of Special Interest (AESI)
Description: AESI Definition:
  The following cluster of symptoms suggestive of CHIKV infection with or without remissions or exacerbations received particular consideration:
  1. Fever (≥38.0°C [100.4°F] measured orally) and
  2. Acute (poly)arthralgia/arthritis most frequently in the extremities (wrists, ankles, and phalanges, often symmetric), back pain and/or neurological symptoms (e.g. confusion, optic neuritis, meningoencephalitis, or polyneuropathy) and/or cardiac symptoms (e.g. myocarditis) or One or more of the following signs and symptoms: macular to maculopapular rash (sometimes with cutaneous pruritus [foot plant] and edema of the face and extremities), polyadenopathies; and
  3. Onset of symptoms 2 to 21 days after vaccination and
  4. Duration of event ≥3 days.
  Ongoing AESIs are monitored for entire study period
Time Frame: within 2 to 21 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 1 | 0

17. Secondary Outcome: Frequency of Any Adverse Event of Special Interest (AESI)
Time Frame: Within 2 to 21 Days Post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
Number analyzed (Participants) | 136 | 137 | 135
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to Month 6
Description: Solicited AEs are collected by systematic assessment through subject eDiaries (within 10 days postvaccination):
  injection site AEs (pain, tenderness, induration, swelling, erythema/redness) or systemic AEs (headache, myalgia, arthralgia, fever, vomiting, nausea, rash, fatigue). Unsolicited AEs, and SAEs are collected by non-systematic assessment up to Day 180.
  AESI is defined as symptoms suggestive of CHIKV infection up to 21 days after vaccination and collected by systematic assessment.
Arm/Group | VLA1553 Lot 1 | VLA1553 Lot 2 | VLA1553 Lot 3
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/137 | 0/135
Serious Adverse Events (participants affected / at risk) | 3/136 | 2/137 | 0/135
Other Adverse Events (participants affected / at risk) | 90/136 | 91/137 | 92/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA1553 Lot 1 (N=136) | VLA1553 Lot 2 (N=137) | VLA1553 Lot 3 (N=135)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA1553 Lot 1 (N=136) | VLA1553 Lot 2 (N=137) | VLA1553 Lot 3 (N=135)
Fatique (General disorders) | 53 (54) | 49 (49) | 55 (56)
Headache (Nervous system disorders) | 49 (56) | 42 (42) | 57 (59)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (34) | 36 (36) | 30 (30)
Injection site pain (General disorders) | 22 (26) | 30 (32) | 22 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (25) | 22 (22) | 26 (31)
Nausea (Gastrointestinal disorders) | 16 (17) | 20 (20) | 17 (17)
Pyrexia (General disorders) | 16 (17) | 18 (18) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) | 6 (7)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (7) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 5 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 5 (5)
Injection site induration (General disorders) | 3 (3) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Injection Site Swelling (General disorders) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (4)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (4) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT04786444/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT04786444/SAP_001.pdf